CLINICAL TRIAL: NCT05449288
Title: Psychometric Properties and Cultural Adaptation of Urdu Version of Modified Oswestry Low Back Pain Scale Among Pakistani Low Back Pain Patients
Brief Title: Urdu Version Of Modified Oswestry Low Back Pain Scale; A Reliability And Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00273
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Radiculopathy
Keywords: Modified Oswestry Low Back Pain Scale; Urdu Version; Reliability; Validity; Lumbar Radiculopathy; Low Back Pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ultimate goal of this study is to interpret Modified Oswestry Low Back Pain Scale into Urdu and analyse its reliability and validity in the population of Pakistan lumber radiculopathy patients. Examine its correlation with Quebec back pain disability scale and the visual analogue scale, as well as the Roland-Morris disability questionnaire.

DETAILED DESCRIPTION:
As per preceding commendation, Modified Oswestry Low Back Pain Scale will be translated into Urdu language from its English version and adapted culturally in Pakistan. 100 individuals will be selected on the basis of convenience sampling with clinical characteristics. The patient will answer the questionnaire package that included the Urdu version Modified Oswestry Low Back Pain Scale, Quebec back pain disability scale, Roland-Morris disability questionnaire and Visual analogue scale on the same day, with a 30-minute delay between the first and second application. Observer-1 will be conducting a third assessment after 7 days for intra-observer evaluation. Statistical Package of Social Sciences Version 24 will be used to enter and evaluate the data. Internal consistency will be measured using the Cronbach alpha value. To evaluated test-retest reliability, an intraclass correlation coefficient will be employed. The Modified Oswestry Low Back Pain Scale will be evaluated for content validity, construct validity, criterion validity, and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, between the ages of 18 to 65,
* Individuals who could read and speak Urdu as a first language
* People who have been diagnosed with lumbar radiculopathy by a physician or neurosurgeon,
* Low Back Pain in the lower extremities with or without radicular pain.

Exclusion Criteria:

* Female patients who were pregnant
* Patients with a mental health history, cancer, or neurological problems
* Acute low back pain is a frequent disease (included recent thoraco-lumbar trauma),
* Psychiatric and behavior issues, systemic disease (tumors and rheumatological diseases), and central or peripheral neurological problems
* Patients who had recently had a cerebrovascular accident or a myocardial infarction were also ruled out.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani Lumber radiculopathy population with low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry Low Back Pain Scale | 1st day
  The Modified Oswestry Low Back Pain Scale includes one item for pain and nine items for daily living activities (personal care, lifting, walking, sitting, standing, sleeping, social life, and travel, employment/homemaking). There are a total of ten items in this scale. Each item is rated on a 6-point ordinal scale, with the best scenario being the best and the worst scenario being the worst.
Quebec back pain disability scale | 1st day
  The Quebec back pain disability scale assesses the degree of functional impairment. The items reflect basic everyday tasks that people with back discomfort may find challenging to do. Bed/rest (items 1-3), sitting/standing (items 4-6), ambulation (items 7-9), mobility (items 10-12), bending/stooping (items 13-16), and handling of large/heavy things (items 17-20) are the six domains of activity impacted by back pain. There are a total of 20 items in this scale.
Roland-Morris disability questionnaire | 1st day
  Roland-Morris disability questionnaire has a total of 24 components. Housework, sleeping, mobility, dressing, obtaining help, eating, irritability, and pain intensity are examples of daily physical activities and functions that may be impacted by Low Back Pain.
Visual analogue scale | 1st day
  The Visual Analogue Scale was created to represent the concept of a fundamental continuity. A Visual Analogue Scale is typically a straight stripe measuring 100 mm long, with word descriptions for each end. The patient draws a line through the spot on the line which they believe best describes their present state. The Visual Analogue Scale score is calculated by calculating in millimeters as from the line's left side to the point marked by that of the patient. It usually ranges from "0" indicating "no pain" to the "10" indicating "worst pain".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No